CLINICAL TRIAL: NCT06813937
Title: Peripheral Magnetic Stimulation (PMS) Effects on Somatosensory Perception in Patients with Upper Limb Amputation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: Motorica LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Skoltech-CNBR6
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Phantom Limb Pain
Keywords: Neuromodulation; Phantom limb pain; Neuropathic pain; Neurostimulation; Chronic pain; Peripheral magnetic stimulation; PMS; Amputation; Amputees
MeSH Terms: conditions — Phantom Limb; Neuralgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Procedure: Peripheral Magnetic Stimulation (PMS) — PMS is a non-invasive neuromodulation technique used to treat chronic pain. Procedure starts with sensory mapping, localisation of the hotspot and detection of sensory threshold. Then two protocols of PMS are implemented: 5 blocks of PMS of varying frequency and 1 block of rPMS.
Other: Electroencephalography (EEG) — EEG is a technique commonly used for the registration of brain activity. The procedure is non-invasive, electrodes are placed on the scalp of the participants. The recording is made simultaneously with the PMS.

SUMMARY:
The study investigates the capabilities of peripheral magnetic stimulation (PMS) as a tool for creating somatosensory sensations of various submodalities and analyzing the dynamics of bioelectric signals of the brain (using encephalography (EEG)) in healthy participants and participants with upper limb amputations. During the experiment, the participants' subjective sensations and EEG activity are recorded in response to magnetic pulses of varying intensity. In addition, the continuous PMS stimulation protocol and its effect on phantom sensations in participants with amputations will be tested for subsequent implementation in clinical practice.

ELIGIBILITY:
For Healthy Volunteers:

Inclusion Criteria:

1. Availability of signed written informed consent.
2. Absence of somatic and psychiatric diseases (more details in the exclusion criteria)
3. Ability and willingness to comply with the requirements of this protocol. Inclusion Criteria

Exclusion Criteria:

1. History of epilepsy (participant, participant's close relatives)
2. Presence of metal or/and electric stimulators and/or implants in participant's body
3. Presence of psychiatric disorders (including a history of), severe depression, suicidal tendencies, or a history of suicide attempts.
4. History of cancer.
5. Complicated traumatic brain injury (TBI) or a history of stroke.
6. Drug addiction (including a history of).
7. Congenital anomaly of upper limb development.
8. Anomalies in the development of the central and peripheral nervous systems.
9. Pregnancy

For stroke patients:

1. History of epilepsy (participant, participant's close relatives)
2. Presence of metal or/and electric stimulators and/or implants in participant's body
3. Presence of psychiatric disorders (including a history of), severe depression, suicidal tendencies, or a history of suicide attempts.
4. History of cancer.
5. Complicated traumatic brain injury (TBI) or a history of stroke.
6. Drug addiction (including a history of).
7. Congenital anomaly of upper limb development.
8. Anomalies in the development of the central and peripheral nervous systems.
9. Pregnancy
10. Presence of severe somatic pathology
11. Presence of severe orthopedic deformity in the limb above the level of amputation.
12. Purulent-septic pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-09-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
1. Visual analogue scale (VAS) | Up to 4 months
  The Visual Analog Scale (VAS) is a 10 cm line used to measure pain intensity. One end of the line represents no pain; while the other end signifies worst possible pain"; The line can be either horizontal or vertical.

SECONDARY OUTCOMES:
Sensory threshold | Up to 6 months
  In this experiment, the goal is to determine the minimum stimulation amplitude that elicits a sensory response. Participants are stimulated by PMS on different power levels and describe their sensations. PMS of the median nerve should evoke tactile response without the muscle response in the area of the palm and fingers which are innervated by it. Sensory threshold is the minimum intensity level which evokes sensory sensations in this particular area.
Sensory mapping | Up to 4 months
  Participants mark their sensations evoked by PMS using PerceptMapper on the scale from 0 (no sensation) to 10 (uncomfortably intense). Participants also mark sensation location on a hand image, describe the sensation's naturalness and intensity and some characteristics of these sensations (tingling, temperature change, et.c.).
Pain detect | Up to 1 year
  The questionnaire combines a pain distribution diagram with a visual analog scale (VAS) and a section focused on identifying spontaneous and triggered neuropathic pain symptoms. It also assesses the nature of pain using the diagram, categorizing it as constant, episodic, or constant with episodes, among others. The questionnaire comprehensively reflects all possible pain parameters, allowing for clear tracking of pain dynamics over time. Its diagnostic accuracy is 83%.
DN4 | Up to 1 year
  The DN4 (Douleur Neuropathique 4) questionnaire is a diagnostic tool designed to identify neuropathic pain, caused by nerve damage. It includes 10 items divided into two sections. The first part consists of seven questions that assess the patient's pain symptoms, such as burning, tingling, electric shocks, or numbness. The second part involves a clinical examination where the physician tests for reduced sensitivity to touch and pinprick, as well as pain response to light brushing. Each item is scored with 1 point for "Yes" and 0 for "No." A total score of 4 or higher indicates a high probability of neuropathic pain.

OTHER OUTCOMES:
Social-demographic questionnaire | Up to 1 year
  Participants fill in the form about their background in their professional sphere and their experience as sportsmen and musicians. This measure can help determine the possible connections between the background and the individual results and enhance personalized care, ultimately leading to better patient outcomes and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Skolkovo Institute of Science and Technology (Skoltech), Moscow, Russia